CLINICAL TRIAL: NCT03505814
Title: Does High Flow Nasal Cannula Oxygen Therapy Prevent Reintubation in Pediatric Surgical Intensive Care Unit
Brief Title: Interest of High Flow Nasal Cannula Oxygen Therapy in Pediatric Intensive Care Unit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hôpital d'enfants Béchir-Hamza (Other)
Responsible Party: Principal Investigator, Dr Sonia ben khalifa (PhD), PROFESSOR, Hôpital d'enfants Béchir-Hamza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HEBechirHamza
Record Dates: First submitted 2018-04-03; First posted 2018-04-23 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Weaning Failure
Keywords: post extubation care; neonatal surgical critical care; oxygen therapy; high nasal flow cannula

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optiflow Group (Experimental): high flow (6l/min), humidified oxygen administred into nasal cannula for post-extubation new born ventilated patients.
  Interventions: Device: High Flow Nasal Cannula Oxygen therapy (OPTIFLOW®)
- Control Group (Active Comparator): Conventional oxygen therapy for post extubation care
  Interventions: Device: Conventional oxygen therapy

INTERVENTIONS:
Device: High Flow Nasal Cannula Oxygen therapy (OPTIFLOW®) — High flow and humidified oxygen support for new borns and young infants for post-extubation care
  Arms: Optiflow Group
Device: Conventional oxygen therapy — conventional oxygen support for new born and young infants in post-extubation care
  Arms: Control Group

SUMMARY:
monocentric randomized controlled trial starting from Mars 2017, recruitment is still ongoing. Patients aged between 0-45 days needing mechanical ventilation (MV) with tracheal intubation were included random assignation in two groups for post-extubation management: Group Optiflow (GO) for patients receiving High Flow Nasal Cannula Oxygen Therapy HNFC and Control Group (CG) for conventional treatment.

Patients were evaluated during the first 72h following extubation. Primary endpoint was the incidence of reintubation. Secondary endpoints were incidence of post-extubation respiratory failure, time to reintubate and weaning time from oxygen. Respiratory and hemodynamic parameters were assessed and compared between the two groups upon extubation, after 2 hours (H2), at H6, H12, H24, H36, H48 and H72. Length of stay (LOS) and mortality were also estimated.

DETAILED DESCRIPTION:
We conducted a monocentric randomized controlled trial starting from Mars 2017, recruitment is still ongoing. Patients aged between 0-45 days needing mechanical ventilation (MV) with tracheal intubation were included regardless type of admission, severity of disease and randomly assigned in two groups for post-extubation management: Group Optiflow (GO) for patients receiving HNFC oxygen therapy and Control Group (CG) for conventional treatment. Before programmed extubation, newborns and young infants received 0.15 mg/kg of Dexamethasone. Patients were evaluated during the first 72h following extubation. Primary endpoint was the incidence of reintubation. Secondary endpoints were incidence of post-extubation respiratory failure, time to reintubate and weaning time from oxygen. Respiratory and hemodynamic parameters were assessed and compared between the two groups upon extubation, after 2 hours (H2), at H6, H12, H24, H36, H48 and H72. Length of stay (LOS) and mortality were also estimated.

ELIGIBILITY:
Inclusion Criteria:

* need for mechanical ventilation
* tracheal intubation
* surgical intensive care admission
* availability of extubation criteria

Exclusion Criteria:

* prior extubation and mechanical ventilation to the actual episode
* weaning failure due to neurological status

Ages: 1 Day to 45 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-08-31 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
reintubation rate | 72 hours following prior weaning and extubation
  need for mechanical ventilation support with tracheal intubation

SECONDARY OUTCOMES:
incidence of post-extubation respiratory failure | 72 hours following prior weaning and extubation
  respiratory failure
time to reintubate | 72 hours following prior weaning and extubation
  time between first extubation and reintubation
weaning time from oxygen. | 72 hours following prior weaning and extubation
  time to wean from any oxygen supply
blood pressure | 72 hours following prior weaning and extubation
  blood pressure
heart rate | 72 hours following prior weaning and extubation
  heart rate
respiratory rate | 72 hours following prior weaning and extubation
  respiratory rate
SpO2/FiO2 | 72 hours following prior weaning and extubation
  pulsed oxygen saturation and inspired fraction of oxygen ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital d'Enfants Bechir Hamza, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided